CLINICAL TRIAL: NCT05230134
Title: Cervical Sympathetic Block to Increase Cerebral Blood Flow in Patients With Cerebral Vasospasm Following Aneurysmal Subarachnoid Hemorrhage
Brief Title: Cervical Sympathetic Block in Patients With Cerebral Vasospasm
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Maria Bombardieri, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64105
Record Dates: First submitted 2022-01-19; First posted 2022-02-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Anesthesia, Local; Cerebral Vasospasm; Subarachnoid Hemorrhage, Aneurysmal
Keywords: regional anesthesia; cervical sympathectomy; cerebral blood flow
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical sympathetic block (Experimental): Patients hospitalized in the ICU and developing clinical manifestations of cerebral vasospasm will be transferred to the neuro-interventional radiology suite for vasospasm treatment. After the vasospasm is confirmed by the angiography followed by a FP-CTP scan, a cervical sympathetic nerve block under ultrasound guidance will be performed. The block consists in the deposition of local anesthetic at the cervical sympathetic ganglion that will be visualized with an ultrasound device. The spread of the local anesthetic will be assessed by performing an 8-second head/neck C-arm CT scan. Another run of angiography and a second FP-CTP will be repeated to check the effect of the block on the brain vasculature after the block is done.
  Patients will have a daily monitoring of their neurological function and of their cerebral blood flow with transcranial doppler in the ICU.
  Interventions: Procedure: Cervical sympathetic block

INTERVENTIONS:
Procedure: Cervical sympathetic block — All participants will get the cervical sympathetic block and catheter under ultrasound guidance.

SUMMARY:
The purposes of this study are twofold: 1) to assess the effect of a cervical sympathetic block on cerebral blood flow in patients suffering from cerebral vasospasm, after aneurysmal subarachnoid hemorrhage; 2) to evaluate the effect of the sympathetic block on the recovery of the neurological function.

DETAILED DESCRIPTION:
Patients hospitalized in the intensive care unit (ICU) and developing clinical manifestations of cerebral vasospasm will be transferred to the neuro-interventional radiology suite for vasospasm treatment. After the vasospasm is confirmed by the angiography followed by a flat panel-computed tomography perfusion (FP-CTP) scan, a cervical sympathetic nerve block under ultrasound guidance will be performed.

The block consists of the deposition of local anesthetic at the cervical sympathetic ganglion that will be visualized with an ultrasound device. The local anesthetic solution with be mixed with a radiographic contrast agent to check the spread of the injectate in the desired anatomical location. The spread of the local anesthetic will be assessed by performing an 8-second head/neck C-arm CT scan. Following the block, another run of angiography and a second FP-CTP will be repeated to assess changes in vessels diameter and in perfusion parameters following the sympathetic block.

Patients will have a daily monitoring of their neurological function and of their cerebral blood flow with transcranial doppler in the ICU.

At 12 months post-aSAH, the patients will complete neurological and neuropsychological assessments as a part of the standard of care. The results of these tests will be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and over
* patients hospitalized in the ICU and developing cerebral vasospasm after aneurysmal subarachnoid hemorrhage

Exclusion Criteria:

- known advanced stage kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | 1 hour after the block
  Cerebral blood flow as measured by computed tomography perfusion
Neurological function | Duration of recovery in ICU (1-2 weeks)
  Change in neurological status as assessed by the Glasgow Coma Scale. The Glasgow Coma Scale score can range from 3 (completely unresponsive) to 15 (responsive).

SECONDARY OUTCOMES:
Cerebral blood flow velocity | Daily during recovery in ICU (1-2 weeks)
  Transcranial doppler measurement
Executive Functioning - Wisconsin Card Sorting Test (WCST) | 12 months post-aSAH
  Measures executive functioning, including cognitive flexibility and problem-solving. The number of categories completed and total errors will be converted to age-adjusted z-scores.
  Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0 (indicative of cognitive impairment in executive functioning).
Processing Speed - Symbol Digit Modalities Test (SDMT) | 12 months post-aSAH
  Assesses visual scanning, tracking, and motor speed. Raw scores are adjusted for age and converted to z-scores. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
Language - Boston Naming Test (BNT) | 12 months post-aSAH
  Evaluates confrontational word retrieval and naming ability. Scores are standardized using age norms. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
Verbal Fluency - FAS Test | 12 months post-aSAH
  Tests lexical fluency by asking participants to generate words beginning with F, A, and S in a set time period. Z-scores are calculated from age-adjusted norms. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
Memory - Hopkins Verbal Learning Test-Revised (HVLT-R) | 12 months post-aSAH
  Assesses verbal learning and memory, including immediate recall, delayed recall, and recognition. Performance is normed and converted into z-scores. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
General mental status - Montreal Cognitive Assessment (MoCA) | 12 months post-aSAH
  Screens for mild cognitive impairment across multiple cognitive domains. Raw scores range from 0 to 30. Favorable outcome: MoCA score ≥ 26, unfavorable outcome: MoCA score < 26 (suggestive of cognitive impairment).
Functional disability - modified Rankin scale (mRS) | 12 months post-aSAH
  Measurement of functional disability using mRS, categorized as favorable (0-3) or unfavorable (4-6), to assess long-term disability and its association with baseline perfusion.
Health-Related Quality of Life (HRQoL, SF-36) | 12 months post-aSAH
  HRQoL will be reported as standardized z-scores, with higher scores indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Bombardieri, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu N, Wu Y, Chen BZ, Han JF, Zhou MT. Protective effect of stellate ganglion block on delayed cerebral vasospasm in an experimental rat model of subarachnoid hemorrhage. Brain Res. 2014 Oct 17;1585:63-71. doi: 10.1016/j.brainres.2014.08.012. Epub 2014 Aug 13. PMID 25128600
- [Background] Dagistan Y, Kilinc E, Balci CN. Cervical sympathectomy modulates the neurogenic inflammatory neuropeptides following experimental subarachnoid hemorrhage in rats. Brain Res. 2019 Nov 1;1722:146366. doi: 10.1016/j.brainres.2019.146366. Epub 2019 Aug 8. PMID 31401069
- [Background] Treggiari MM, Romand JA, Martin JB, Reverdin A, Rufenacht DA, de Tribolet N. Cervical sympathetic block to reverse delayed ischemic neurological deficits after aneurysmal subarachnoid hemorrhage. Stroke. 2003 Apr;34(4):961-7. doi: 10.1161/01.STR.0000060893.72098.80. Epub 2003 Mar 20. PMID 12649526
- [Background] Zhang J, Nie Y, Pang Q, Zhang X, Wang Q, Tang J. Effects of stellate ganglion block on early brain injury in patients with subarachnoid hemorrhage: a randomised control trial. BMC Anesthesiol. 2021 Jan 20;21(1):23. doi: 10.1186/s12871-020-01215-3. PMID 33472582
- [Background] Pileggi M, Mosimann PJ, Isalberti M, Piechowiak EI, Merlani P, Reinert M, Cianfoni A. Stellate ganglion block combined with intra-arterial treatment: a "one-stop shop" for cerebral vasospasm after aneurysmal subarachnoid hemorrhage-a pilot study. Neuroradiology. 2021 Oct;63(10):1701-1708. doi: 10.1007/s00234-021-02689-9. Epub 2021 Mar 16. PMID 33725155